CLINICAL TRIAL: NCT05997810
Title: A Phase 2 Biomarker Study of Parathyroid Tumor Clonal Status in Primary Hyperparathyroidism
Brief Title: Parathyroid Tumor Clonal Status
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202212100
Record Dates: First submitted 2023-08-04; First posted 2023-08-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Parathyroid Tumor; Primary Hyperparathyroidism
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen samples will be obtained from FFPE tumor slides, Fresh-frozen tissue, and Blood.
  NOTE: Fresh-frozen tumor, normal gland biopsy and blood samples will be collected at the WUSM study site only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To define the frequency of monoclonal-X and polyclonal-X tumors in PHPT participants having parathyroidectomy (PTX) and to define the relationship between parathyroid tumor clonal status and multiple gland neoplasia (MGN), we will compare surgical and pathologic outcomes to tumor clonal status in a multicenter cohort of patients having bilateral neck exploration (BNE) and PTX (primary objectives).

DETAILED DESCRIPTION:
To define the frequency of monoclonal-X and polyclonal-X tumors in primary hyperparathyroidism (PHPT) participants having parathyroidectomy (PTX) and to define the relationship between parathyroid tumor clonal status and multiple gland neoplasia (MGN), the investigators will compare surgical and pathologic outcomes to tumor clonal status in a multicenter cohort of participants having bilateral neck exploration (BNE) and PTX.

Study participants will be recruited from four high-volume centers at Washington University in St. Louis (WU), University of California San Francisco, University of Alabama-Birmingham, and the University of Pennsylvania. Eligible participants will receive standard of care treatment (parathyroidectomy) and de-identified formalin-fixed paraffin-embedded (FFPE) tumor samples (stained and unstained from each abnormal gland) will be sent to WU for study. DNA will be extracted from FFPE samples and the HUMARA assay will be performed according to our established protocol. Our two published studies show >90% concordance between replicate HUMARA assays of the same tumor. For additional rigor, two regions of each tumor will be assayed independently to ensure concordance of clonal status. Tumors where the clonality call from the two within-tumor samples are discordant will be recorded as such, and the investigators will perform sensitivity analyses, for aims where this is relevant, of assigning one or the other clonal state to these samples.

Further, the investigators will employ a secondary assay (Cytoscan HD array, ThermoFisher) to assess DNA copy number variation (CNV) in a random set of samples from 58 polyclonal-X cases and 49 monoclonal-X cases (estimated 107 total assays). Published and unpublished data have shown that CNV occurs with considerable frequency in parathyroid tumors, including adenomas. CNV assessment can provide independent verification of an X-inactivation-based finding of polyclonality by identifying heterogeneous CNV within a tumor sample indicating polyclonality, or more uniform CNV reflecting monoclonality. Cases with discordant results (estimated <10%) from HUMARA and CNV assays will be comprehensively studied in the exploratory objectives.

De-identified pathologic data including the number and weight of abnormal glands removed from participants will be recorded at local study sites and entered in a REDCap database maintained at WU. The Investigators then will review operative and pathologic reports for correlation of tumor clonality and the presence of single gland neoplasia (SGN) or multiple gland neoplasia (MGN). In cases of MGN the investigators will perform ms-PCR of HUMARA alleles on all resected tumors to assess for concordance of clonality. The investigators will also determine the impact of two common surgical approaches on outcomes in tumors of different clonal status. The frequency of MGN stratified by tumor clonality will be examined in participants who undergo UNE with ioPTH monitoring and compared BNE. Operative and pathology reports will be reviewed as well as ioPTH levels drawn before and both 5 and 10 minutes (PTH T1/2 = 5 min.) after tumor removal. Underlying tumor clonality will be determined as described above and will be compared to pathologic results (MGN versus SGN), as well as ioPTH kinetics (% decline from pre-op PTH levels at 5 and 10 minutes after final tumor removal).

To define the relationship between parathyroid tumor clonal status and biochemical outcomes following PTX for PHPT, the investigators will compare baseline clinical features, surgical/pathologic findings and postoperative biochemical outcomes following PTX to tumor clonal status in a large, multicenter cohort of participants having PTX. A total of 645 participants with known tumor clonal status will have standard clinical and biochemical data (serum calcium, albumin, intact PTH, 25(OH)D, and creatinine) recorded at baseline (before PTX), and at 2 weeks, 3 months, and 6 months post-PTX (not all labs are recorded at each follow-up time point). The investigators will compare the frequency of elevated PTH (ePTH) at each time point in participants with monoclonal-X and polyclonal-X tumors. The investigators have previously shown that vitamin D status impacts ePTH following PTX. To investigate abnormal vitamin D metabolism, the most common mechanism of secondary hyperparathyroidism as a cause of polyclonal-X disease, the investigators also will perform a comprehensive analysis of vitamin D status in a subset of 111 WUSM participants with monoclonal-X and polyclonal-X tumors. Our analysis will include biochemical indices of vitamin D metabolism (25-hydroxyvitamin D, 1,25-dihydroxyvitamin D and vitamin D binding protein levels).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with nonfamilial primary hyperparathyroidism biochemically confirmed by measurement of serum calcium and intact PTH within 60 days of enrollment.
* Female.
* Age ≥ 18 years
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Patients with a history of cervicofacial irradiation.
* Patients with recurrent or persistent PHPT after prior PTX.
* Patients with secondary hyperparathyroidism due to renal failure on renal replacement therapy (i.e. hemodialysis or peritoneal dialysis).
* Patients with tertiary hyperparathyroidism due to renal failure with or without history of renal transplantation.
* Patients receiving calcimimetic agents (e.g. cinacalcet / Sensipar) within 30 days of PTX.
* Patients currently taking lithium or with a history of lithium use.
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females scheduled to have surgery for primary hyperparathyroidism.
Sampling Method: Non-Probability Sample
Enrollment: 839 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint 1 | 24 months
  Frequency of occurrence of monoclonal-X versus polyclonal-X parathyroid tumors in a prospective multi-center cohort of patients having parathyroidectomy for primary hyperparathyroidism.
Primary Endpoint 2 | 24 months
  Determine clinicopathologic features of monoclonal-X versus polyclonal-X parathyroid tumors in a prospective multi-center cohort of patients with PHPT referred for PTX.
Primary Endpoint 3 | 24 months
  Perform a prospective study of biochemical outcomes of PTX in PHPT patients with monoclonal-X and polyclonal-X tumors.

SECONDARY OUTCOMES:
Secondary Endpoint | 24 months
  To investigate mechanism(s) of monoclonal-X and polyclonal-X parathyroid tumorigenesis using functional and genomic approaches (e.g. calcium sensing capacity determined by EC50 and single nucleotide variants / copy number variation).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - University of California-Department of Surgery, San Francisco, California
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania